CLINICAL TRIAL: NCT00304824
Title: Olfactory Function in Glaucoma Patients
Brief Title: Assessment of the Ability to Distinguish Odors in Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgül, MD, University Hospital, Basel, Switzerland
Other Study IDs: 009-Guk-2004-002
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Olfactory functions; Sniffing Sticks Test
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glaucoma is one of the leading causes of blindness worldwide. The key feature of glaucoma is damage to the optic nerve head with loss of retinal ganglion cells and local tissue remodeling. Neuronal cell death in glaucoma occurs by apoptotic mechanisms1. Apoptosis of neurons also plays a major role in neurodegenerative diseases, such as Alzheimer's or Parkinson's disease. An association between glaucoma and these disorders has been described 2-4. Furthermore, it has been reported that the olfactory function is disturbed in these neurodegenerative diseases5-6. We hypothesize that similar olfactory alterations may occur in glaucoma which is in fact a local neurodegenerative disease.

DETAILED DESCRIPTION:
1. Introduction

   1. Background and rationale of the study Glaucoma is one of the leading causes of blindness worldwide. The key feature of glaucoma is damage to the optic nerve head with loss of retinal ganglion cells and local tissue remodeling. Neuronal cell death in glaucoma occurs by apoptotic mechanisms1. Apoptosis of neurons also plays a major role in neurodegenerative diseases, such as Alzheimer's or Parkinson's disease. An association between glaucoma and these disorders has been described 2-4. Furthermore, it has been reported that the olfactory function is disturbed in these neurodegenerative diseases5-6. We hypothesize that similar olfactory alterations may occur in glaucoma which is in fact a local neurodegenerative disease.
   2. Study objectives Primary Objective: To test the olfactory function in glaucoma patients.
   3. Investigational plan Chronic glaucoma patients will be assessed regarding inclusion/exclusion criteria and clinical criteria. A basic otorhinolaryngological examination addressing the possible exclusion criteria will be performed prior to the Sniffing Sticks test battery. A simple questionnaire regarding an olfactory status of the patient will be filled out. The olfactory performance of glaucoma patients will be compared to the existing age-matched normative database.
   4. Design Single center cohort study, normative database as control.
   5. Selection of study population

      I. Number of subjects Thirty consecutive glaucoma patients, age 18 - 70, will be recruited from the glaucoma consultation at the University Eye Clinic Basel.

      II. Prestudy screening A detailed medical and ophthalmic history will be recorded and all patients will complete an ophthalmologic examination (best corrected visual acuity, intraocular pressure measurements, slit-lamp examination, indirect fundoscopy) as well as an otorhinolaryngological examination.

      III. Inclusion criteria Diagnosis of chronic open-angle glaucoma will be based on the presence of typical glaucomatous disc damage and visual field defects. Only patients with a recent gonioscopic examination and at least two visual field examinations will be recruited.

      IV. Exclusion criteria Occludable iridocorneal angles, a history of current, chronic or recurrent inflammatory eye disease, a history of retinal or neuroophthalmologic disease that could result in visual field defects, need for any concomitant medications that may interfere with the evaluation of olfactory function, a history of past or active alcohol or drug abuse, smoking, a history of olfactory disturbance related to identifiable local factors, and any local condition that could lead to hyposmia/anosmia or interfere with the olfactory function, such as polyps, chronic sinus infection, sub(acute) viral or bacterial infection, history of sinus surgery, will be considered as an exclusion criterion.

      V. Study medication NA
   6. Study protocol I. General restrictions on subjects NA

      II. Dietary restriction NA.

      III. Description of study days On the experimental day a detailed history will be taken and a complete ophthalmologic examination including best corrected visual acuity, slit-lamp examination, indirect fundoscopy, and intraocular pressure measurement will be performed (KG). Based on these examinations and chart data, the patient shall be classified as glaucoma patient. A basic otorhinolaryngological screening examination will follow, the patient will fill an olfactory questionnaire and the Sniffing Sticks test battery will be performed (AWL).
   7. Efficacy variables I. Outcome variables Odor threshold score (0-16), odor discrimination task score (0-16), Odor identification score (0-16), composite score (sum of the three above).

   II. Follow-up safety investigations NA
2. Methods of evaluation

   a. Sniffing Sticks test battery7 Commercially available felt-tip pens, 14 cm long and with an inner diameter of 1.3 cm, are filled with 4 mL of liquid odorants or odorants dissolved in propylene glycol. For odor presentation the cap is removed by the experimenter for approximately 3 seconds and the pen's tip is placed 2 cm in front of the examined nostril. Three tests are performed. Odor threshold for n-butanol is assessed using a single-staircase, triple-forced choice procedure. Sixteen dilutions are prepared. Three pens are presented at randomized order, with two containing only the solvent. The patient's task is to identify the odor-containing pen. The score ranges from 0 to 16. In the odor-discrimination test, the patient has to determine which of the three presented pens smell differently. A total of 16 triplets is presented to the patient, and thus the score ranges from 0 to 16. Odor identification is assessed by means of 16 common odors, using a multiple choice technique with a list of four descriptors. The score ranges also from 0 to 16. The composite score is the sum of three scores.
3. Statistical procedures

   1. Biometric methods Mann-Whitney U-test, p<0.05 being considered significant.
   2. Statistical model Olfactory scores of glaucoma patients will be compared to the age-matched normative database by means of Mann-Whitney U-test.
   3. Study power No power calculations were performed, as there are no prior pilot studies.

ELIGIBILITY:
Inclusion Criteria:

Chronic open-angle glaucoma with typical glaucomatous disc and visual field damage.

Exclusion Criteria:

* Occludable iridocorneal angles
* History of current, chronic or recurrent inflammatory eye disease
* History of retinal or neuroophthalmologic disease that could result in visual field defects
* Need for any concomitant medications that may interfere with the evaluation of olfactory function
* Patients with a significant history and/or active alcohol or drug abuse (significant is defined as that which in the opinion of the investigator may either put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study), smokers
* History of olfactory disturbance related to identifiable local factors and any local condition that could lead to hyposmia/anosmia or interfere with the olfactory function, such as polyps, chronic sinus infection, sub(acute) viral or bacterial infection, history of sinus surgery

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-10; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgul, Study Director — University Eye Hospital Basel, Switzerland

REFERENCES:
- See also: University Basel, Switzerland — http://www.unibas.ch